CLINICAL TRIAL: NCT06322745
Title: Thulium Beam Coagulation Versus Suture Renorrhaphy for Hemostasis of Tumor Bed in Laparoscopic Partial Nephrectomy: Prospective Randomized Comparative Study
Brief Title: Thulium Beam Coagulation Versus Suture Renorrhaphy for Hemostasis of Tumor Bed in Laparoscopic Partial Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Mohammed Ali Atallah, Assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1986
Record Dates: First submitted 2024-03-07; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Renal Tumor; Renal Malignant Tumor
Keywords: Thulium laser; Laparoscopic partial nephrectomy; Ischemia time; Small renal mass
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: A randomized prospective comparative study. Two-arm parallel assignment:
  First Arm: involves cases of laparoscopic partial nephrectomy done with suture renorrhaphy only for hemostasis of the tumor bed.
  Second Arm: involves cases of laparoscopic partial nephrectomy using thulium beam coagulation and suture renorrhaphy for hemostasis of the tumor bed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suture renorrhaphy group (Active Comparator): involves cases of laparoscopic partial nephrectomy done with suture renorrhaphy only for hemostasis of the tumor bed.
  Interventions: Procedure: Suture renorrhaphy only for hemostasis of the tumor bed in laparoscopic partial nephrectomy
- thulium beam coagulation group (Active Comparator): involves cases of laparoscopic partial nephrectomy with thulium beam coagulation and suture renorrhaphy for hemostasis of the tumor bed
  Interventions: Procedure: Thulium beam coagulation and suture renorrhaphy for hemostasis of the tumor bed in laparoscopic partial nephrectomy

INTERVENTIONS:
Procedure: Suture renorrhaphy only for hemostasis of the tumor bed in laparoscopic partial nephrectomy — Suture renorrhaphy will be used in 2 layers; medullary and cortical, with Vicry 2/0 or 3/0 and secured with V-lock. Early unclamping will be done after hemostasis of the medullary layer. Renorrhaphy of the cortical layer will be continued after that.
  Arms: suture renorrhaphy group
Procedure: Thulium beam coagulation and suture renorrhaphy for hemostasis of the tumor bed in laparoscopic partial nephrectomy — A 2-μm continuous thulium laser with 365 μm laser fiber at 30-40 W will be used for coagulation of the tumor bed. Large vessels that may not be completely sealed with thulium beam will be closed by V-lock to achieve safe and stable hemostasis. Early unclamping will be done after hemostasis of the tumor bed. Suture renorrhaphy will be used in 1 layer to approximate the renal parenchyma.
  Arms: thulium beam coagulation group

SUMMARY:
To compare the outcome of thulium beam coagulation versus suture renorrhaphy for hemostasis of the tumor bed in laparoscopic partial nephrectomy.

DETAILED DESCRIPTION:
To date, no studies have compared the outcomes of thulium beam coagulation versus suture renorrhaphy for hemostasis of tumor bed in laparoscopic partial nephrectomy in patients with small renal messes (SRMs).

This study aims to compare the outcome of thulium beam coagulation versus suture renorrhaphy for hemostasis of the tumor bed in laparoscopic partial nephrectomy.

The investigators hypothesize that:

Conducted well designed, randomized prospective comparative study can help to identify which technique is better.

Using thulium beam coagulation for hemostasis of the tumor bed in laparoscopic partial nephrectomy can improve the outcome, shorten intraoperative ischemia time and decrease blood loss.

ELIGIBILITY:
Inclusion Criteria:

* cT1 single renal mass.

Exclusion Criteria:

1. Absolute contraindication for laparoscopic surgery (e.g., severe cardiopulmonary insufficiency, and chronic obstructive lung disease).
2. Renal mass involving the hilum.
3. Renal mass in patients with chronic kidney disease.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Warm Ischemia time (WIT) in minutes (time of renal artery clamping). | during the surgery
  Started once renal artery clamped before tumor enucleation till release of the clamp after 1st layer renorraphy in group 1 or Thulium beam coagulation in group 2
Suture time and operative time in minutes | during the surgery
  Suture time starts from the first suture to the last one, including time of manipulating needles.
Intraoperative number of sutures for renorraphy | during the surgery
  which is the count of each time the needle comes out from the renal parenchyma.
Intraoperative Blood loss | during the surgery
  Blood loss will be calculated from the suction jar minus the amount of fluid irrigation
Blood transfusion rate | perioperatively
  Amount of blood in ml transfused intraoperative or postoperative
Renal function: serum creatinine | 3 months
  will be estimated by serum creatinine. Chronic kidney disease (CKD): will be staged according to Kidney Disease Improving Global Outcomes (KDIGO) guidelines to reflect the change of renal function
Renal function: estimated GFR (eGFR) | 3 months
  ill be estimated by estimated GFR (eGFR) using Modification of Diet in Renal Disease (MDRD) equation (Levey et al., 2006).
  Chronic kidney disease (CKD): will be staged according to Kidney Disease Improving Global Outcomes (KDIGO) guidelines to reflect the change of renal function
Transforming growth factor beta (TGF-β) urine level | pre-surgery, at 24 hours and at 1 month
  will be measured in urine to indicate the fibrogenic process that occurs in renal parenchyma after PN
Monocyte chemoattractant protein (MCP-1) urine level | pre-surgery, at 24 hours and at 1 month
  will be measured in urine to indicate the fibrogenic process that occurs in renal parenchyma after PN

SECONDARY OUTCOMES:
Hospital stay | perioperatively
  from time of surgery till time of patient discharge.
Post operative pain | perioperatively
  by Visual Analogue Scale The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 100 mm line that represents a continuum between "0 or no pain" and "100 or worst pain".

CONTACTS AND LOCATIONS:
Overall Officials: Aly Abdel-Karim, Professor, Study Director — Alexandria University; Abdel-Rahman Ebeid, Professor, Study Director — Al-Azhar University-Cairo
Locations (1):
- Urology Department, Al-Azhar University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Patient data sheet, patient consent forms through my e-mail: Ehab44ehab@gmail.com
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available after 1 year may extend to another 1 year.
Access Criteria: My e-mail: Ehab44ehab@gmail.com